CLINICAL TRIAL: NCT06230289
Title: Effect of 4 Point TAP Block on Diaphragm Thickness in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Transversus Abdominis Plane Block on Diaphragm Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Nuran Akıncı Ekinci, Medical Doctor, Konya City Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DiaTap
Record Dates: First submitted 2023-12-21; First posted 2024-01-30 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Diaphragm; Relaxation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B: Transabdominal plane block group (Active Comparator): Patients agreeing to participate will be allocated to the control group (Group C, n=25) or the block group (Group B, n=25). The allocation will be randomized using a web-based data entry and randomization platform (by using envelope selection method) by an anesthesiologist not involved in the study. At the end of the surgery, patients in Group B will receive a four-point TAP block.
  Interventions: Procedure: Transabdominal plane block
- Group C: Control group with multi-modal analgesia (No Intervention): Patients agreeing to participate will be allocated to the control group (Group C, n=25) or the block group (Group B, n=25). The allocation will be randomized using a web-based data entry and randomization platform (by using envelope selection method) by an anesthesiologist not involved in the study. At the end of the surgery, patients in Group C which will be performed no interventional procedures.

INTERVENTIONS:
Procedure: Transabdominal plane block — Patients agreeing to participate will be allocated to the control group (Group C, n=25) or the block group (Group B, n=25). The allocation will be randomized using a web-based data entry and randomization platform (by using envelope selection method) by an anesthesiologist not involved in the study. At the end of the surgery, patients in Group B will receive a four-point TAP block, while no interventional procedures will be performed on patients in Group C.
  Arms: Group B: Transabdominal plane block group

SUMMARY:
Hypothesis: Postoperative pain, by preventing effective diaphragmatic contraction, hinders deep inspiration and expiration. Inspiratory and expiratory levels can be assessed by measuring diaphragm thickness using ultrasound.Diaphragm thickness[DT] measured at the end of inspiration and expiration will differ between patients who undergo Transversus Abdominis Plane Block[TAP] block using the 4-point technique and those who do not. It is anticipated that in patients who receive the block, diaphragm thickness will be greater, serving as an indicator of

DETAILED DESCRIPTION:
Postoperative pain is among the main reasons for the decrease in respiratory function after upper abdominal surgery. Numerous studies have investigated the relationship between pain and respiratory function in abdominal surgeries. While the classic TAP block is used to relieve lower abdominal pain [Th10-Th12] after surgery, it may be insufficient in relieving pain in the upper abdominal wall [Th6-Th9]. The 4-point TAPb technique is employed to address the pain in this region. Ultrasound allows for non-invasive assessment of changes in diaphragm thickness along with changes in lung volume, and evaluating diaphragm mass and contraction is highly useful in diagnosing respiratory diseases. Previous studies have explored changes in diaphragm thickness and the relationship between total lung capacity [TLC], functional residual capacity [FRC], residual volume [RV] and diaphragm function. However, changes in diaphragm function due to pain prevention in patients undergoing '4-point' TAPb are not well understood. It is aimed to investigate the impact of the 4-point TAP block on the diaphragm in patients undergoing laparoscopic cholecystectomy under general anesthesia. The primary objective of this study is to use ultrasound to examine the effect of the four-point TAP block, administered for analgesia after laparoscopic cholecystectomy, on diaphragm thickness. The secondary objective is to assess the impact of the four-point TAP block on pain and the quality of patient recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. 18-65 years old;
3. ASA Physical Status 1-2;
4. Scheduled for elective kolesistektomi.

Exclusion Criteria:

1. ≤18, ≥65 years old;
2. Any contraindications nerve blocks;
3. VKİ>35 kg/m2;
4. Bleeding diathesis;
5. Switching to open surgery;
6. Language barrier;
7. Having undergone upper abdominal surgery previously;
8. Severe kind of chronic lung ilness;
9. Contraindication or allergy to planned drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Diaphragma thickness as milimeter | Preoperative measurement of DT and postoperative measurement of DT(5. minutes and 30. minutes)
  Measurement of Diaphragm Thickness: Patients will be placed in a supine position with the head elevated 30 degrees, and high-frequency linear probe ultrasound (DC-60 Diagnostic Ultrasound, Shenzhen Mindray, China) will be used to visualize the diaphragm in its characteristic three-layered appearance above the anterior axillary line at the aponeurosis region (lung-pleura). The hypoechoic (dark) muscle tissue between the two hyperechoic (bright) lines of pleural and peritoneal fascia will be imaged, and the thickness will be measured and recorded.

SECONDARY OUTCOMES:
Visual Analog Scale (from 1 to 10) | VAS assessment preoperatively and postoperatively at 5 minutes, 30 minutes, 2 hours, 8 hours, and 24 hours.
  Secondary outcome measures will include preoperative and postoperative assessments at 5 minutes, 30 minutes, 2 hours, 8 hours, and 24 hours, using the Visual Analog Scale (VAS) to evaluate pain for both resting and movement (0-10, 0 = no pain, 10 = the most severe pain).
Opioid consumption as miligram per day | 2, 8, and 24 hours postoperatively assessments
  Secondary outcome measures include preoperative, 5 minutes post-extubation, 30 minutes post-extubation, and 2, 8, and 24 hours postoperatively assessments of total tramadol consumption, the number of patients requiring postoperative rescue analgesia, nausea, vomiting.
Quality of Recovery-15T score (from 0 to150) | 24 hours postoperatively assessments
  Secondary outcome measures include 24 hours postoperatively assessments of the patient recovery score evaluated with QoR-15T will also be recorded. Results: The QoR-15 scores for Excellent: 136-150, Good:122-135, Moderate:90-121, Poor recovery: 0-89.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran Akıncı, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Nuran Akıncı, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After performing the study, we might share all info with the system.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We want to describe the time frame after finish the study as completed.
Access Criteria: We can share the data by using e-mail.